CLINICAL TRIAL: NCT03207893
Title: Benefits of Adding Continuous Glucose Monitoring to Glycemic Load, Exercise, and Monitoring of Blood Glucose (GEM) for Adults With Type 2 Diabetes - Phase 2
Brief Title: Benefits of Continuous Glucose Monitoring With GEM Lifestyle Modification for Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Cox, PhD, Professor, Departments of Psychiatry, Internal Medicine and Ophthalmology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19313
Record Dates: First submitted 2016-10-28; First posted 2017-07-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEM+CGM (Experimental): GEM lifestyle modification & continuous glucose monitoring
  Interventions: Behavioral: GEM lifestyle modification & continuous glucose monitoring; Other: Routine Care
- Routine Care (Active Comparator): Subject's current t2d treatment
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: GEM lifestyle modification & continuous glucose monitoring — Four treatment sessions of GEM lifestyle modification in 3 months and continuous glucose monitoring during the first 14 days of each of the 3 months.
  Arms: GEM+CGM
Other: Routine Care — Subject's current t2d treatment

SUMMARY:
The purpose of this study is to determine if the use of continuous glucose monitoring with the GEM lifestyle modification program (Glycemic load, Exercise and Monitoring glucose) will result in better diabetes control than routine care.

DETAILED DESCRIPTION:
Type 2 diabetes (t2d) is a major epidemic of the developing world which has huge fiscal consequences and many physical complications. It is thought to be brought on in part by contemporary easy access to high energy foods and reduced physical activity, resulting in increased belly fat that culminates in growing insulin resistance and subsequent hyperglycemia. Because of ease and efficacy of medication management, t2d is primarily managed with ever-escalating medication use, which significantly contributes to medical cost and possibly the progression of the disease itself.

An effective supplement or alternative to medication management is lifestyle modification. Conventional lifestyle modification focuses on reducing body fat and insulin resistance through weight reduction from caloric restriction and aerobic exercise. Sustained routine application of this approach is limited because some individuals do not need to lose weight, some do not want to lose weight, others cannot lose weight, and when successful, lifelong weight reduction is difficult to sustain. A useful paradigm shift in lifestyle treatment of t2d might be to go from reducing calories to reducing postprandial glucose (PPG), the primary contributor to glycosylated hemoglobin (HbA1c).

PPG spikes can be prevented by replacing high with low glycemic load foods and dampened by engaging in postprandial physical activity. This is exemplified by the integrated Glycemic load, Exercise and Monitoring glucose (GEM) program. It promotes choices of low glycemic load foods and increased physical activity, directed by glucose monitoring feedback. Glucose feedback can: 1) educate people as to what food choices minimize PPG and what physical activity choices directly lower PPG, 2) activate individuals when glucose is out of their desired range by alerting them to make choices to lower high glucose or raise low glucose, and 3) motivate individuals to repeat those choices that resulted in desirable glucose consequences. The educating, activating and motivating benefits of glucose feedback are thought to be qualitatively and quantitatively enhanced through continuous glucose monitoring (CGM).

It is hypothesized that, compared to Routine Care (RC), GEM with CGM (GEM+CGM) administered to adults with t2d who are failing with oral medication management will result in better diabetes control (lower HbA1c), reduced medication management (less medication), and better psychological functioning (e.g. greater sense of empowerment) in the short term (3 month follow-up). Further, it is hypothesized that their reduction in HbA1c will be driven by a reduction in PPG.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Between the ages of 21 and 80
* Failed on an oral medication regimen (HbA1c > 7.5%).

Exclusion Criteria:

* Takes insulin
* Took medications in the last 3 months that impede weight loss (e.g., prednisone)
* Pregnant or contemplating pregnancy in the next 12 months
* Conditions that preclude increasing physical activity (e.g. severe neuropathy, cardiovascular disease, chronic obstructive pulmonary disease/emphysema, osteoarthritis, stroke)
* Severe mental disease (e.g. manic depressive illness, severe depression, or active substance abuse)
* Undergoing treatment for cancer
* History of lactic acidosis
* Marked renal impairment (eGFR < 45; stage 3b chronic kidney disease)
* Takes psychotropic medications that raise blood glucose (e.g. atypical antipsychotics)
* Cannot read English.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
HbA1c | baseline, 3 months post-intervention
  Change in HbA1c measured via blood test
Medication changes | baseline, 3 months post-intervention
  Changes in prescribed medications (type and/or dosage)

SECONDARY OUTCOMES:
change in food choices (ASA24 survey) | baseline, 3 months post-intervention
  ASA24 survey across 3 separate days
change in food choices (energy bar selection) | baseline, 3 months post-intervention
  At assessment visits, subjects will choose between energy bars that do or dont support the intervention principles.
Exercise (Fitbit) | baseline, 3 months post-intervention
  daily activity will be recorded
change in psychological functioning (dietary habits questionnaire) | baseline, 3 months post-intervention
  The Food Questionnaire
change in psychological functioning (quality of life questionnaire) | baseline, 3 months post-intervention
  WHOQO-BREF Questionnaire
change in psychological functioning (depression questionnaire) | baseline, 3 months post-intervention
  Patient Health Questionnaire (PHQ-9)
change in psychological functioning (numeracy questionnaire) | baseline, 3 months post-intervention
  Numeracy Scale - measures how good one is with numbers
change in psychological functioning (diabetes knowledge questionnaire) | baseline, 3 months post-intervention
  Diabetes Knowledge Scale - measures diabetes knowledge
change in psychological functioning (empowerment questionnaire) | baseline, 3 months post-intervention
  Diabetes Empowerment Scale
Psychological functioning (PAID questionnaire) | baseline, 3 months post-intervention
  Problem Area In Diabetes scale (PAID) - measures concerns about diabetes
change in psychological functioning (attitude towards glucose monitoring questionnaire) | baseline, 3 months post-intervention
  The Glucose Monitoring Satisfaction Survey (GMSS)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Dept. of Psychiatry and Neurobehavioral Sciences, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Cox DJ, Gill Taylor A, Dunning ES, Winston MC, Luk Van IL, McCall A, Singh H, Yancy WS Jr. Impact of behavioral interventions in the management of adults with type 2 diabetes mellitus. Curr Diab Rep. 2013 Dec;13(6):860-8. doi: 10.1007/s11892-013-0423-7. PMID 24072477
- [Background] Hill JO, Galloway JM, Goley A, Marrero DG, Minners R, Montgomery B, Peterson GE, Ratner RE, Sanchez E, Aroda VR. Scientific statement: Socioecological determinants of prediabetes and type 2 diabetes. Diabetes Care. 2013 Aug;36(8):2430-9. doi: 10.2337/dc13-1161. Epub 2013 Jun 20. No abstract available. PMID 23788649
- [Background] Whiting DR, Guariguata L, Weil C, Shaw J. IDF diabetes atlas: global estimates of the prevalence of diabetes for 2011 and 2030. Diabetes Res Clin Pract. 2011 Dec;94(3):311-21. doi: 10.1016/j.diabres.2011.10.029. Epub 2011 Nov 12. PMID 22079683
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] Turner RC, Cull CA, Frighi V, Holman RR. Glycemic control with diet, sulfonylurea, metformin, or insulin in patients with type 2 diabetes mellitus: progressive requirement for multiple therapies (UKPDS 49). UK Prospective Diabetes Study (UKPDS) Group. JAMA. 1999 Jun 2;281(21):2005-12. doi: 10.1001/jama.281.21.2005. PMID 10359389
- [Background] Ceriello A, Davidson J, Hanefeld M, Leiter L, Monnier L, Owens D, Tajima N, Tuomilehto J; International Prandial Glucose Regulation Study Group. Postprandial hyperglycaemia and cardiovascular complications of diabetes: an update. Nutr Metab Cardiovasc Dis. 2006 Oct;16(7):453-6. doi: 10.1016/j.numecd.2006.05.006. Epub 2006 Aug 24. PMID 16934443
- [Background] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] Look AHEAD Research Group; Pi-Sunyer X, Blackburn G, Brancati FL, Bray GA, Bright R, Clark JM, Curtis JM, Espeland MA, Foreyt JP, Graves K, Haffner SM, Harrison B, Hill JO, Horton ES, Jakicic J, Jeffery RW, Johnson KC, Kahn S, Kelley DE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montgomery B, Nathan DM, Patricio J, Peters A, Redmon JB, Reeves RS, Ryan DH, Safford M, Van Dorsten B, Wadden TA, Wagenknecht L, Wesche-Thobaben J, Wing RR, Yanovski SZ. Reduction in weight and cardiovascular disease risk factors in individuals with type 2 diabetes: one-year results of the look AHEAD trial. Diabetes Care. 2007 Jun;30(6):1374-83. doi: 10.2337/dc07-0048. Epub 2007 Mar 15. PMID 17363746
- [Background] DiPietro L, Gribok A, Stevens MS, Hamm LF, Rumpler W. Three 15-min bouts of moderate postmeal walking significantly improves 24-h glycemic control in older people at risk for impaired glucose tolerance. Diabetes Care. 2013 Oct;36(10):3262-8. doi: 10.2337/dc13-0084. Epub 2013 Jun 11. PMID 23761134
- [Background] Mayer-Davis EJ, D'Agostino R Jr, Karter AJ, Haffner SM, Rewers MJ, Saad M, Bergman RN. Intensity and amount of physical activity in relation to insulin sensitivity: the Insulin Resistance Atherosclerosis Study. JAMA. 1998 Mar 4;279(9):669-74. doi: 10.1001/jama.279.9.669. PMID 9496984
- [Background] Ingersoll KS, Banton T, Gorlin E, Vajda K, Singh H, Peterson N, Gonder-Frederick L, Cox DJ. Motivational Interviewing Support for a Behavioral Health Internet Intervention for Drivers with Type 1 Diabetes. Internet Interv. 2015 May 1;2(2):103-109. doi: 10.1016/j.invent.2015.02.001. PMID 25774342
- [Background] Hostmark AT, Ekeland GS, Beckstrom AC, Meen HD. Postprandial light physical activity blunts the blood glucose increase. Prev Med. 2006 May;42(5):369-71. doi: 10.1016/j.ypmed.2005.10.001. Epub 2006 Mar 20. PMID 16549107
- [Background] Robertson RP, Harmon J, Tran PO, Tanaka Y, Takahashi H. Glucose toxicity in beta-cells: type 2 diabetes, good radicals gone bad, and the glutathione connection. Diabetes. 2003 Mar;52(3):581-7. doi: 10.2337/diabetes.52.3.581. PMID 12606496
- [Background] Heinemann L. (Analytical) accuracy of blood glucose meters and patients: how do they come together? J Diabetes Sci Technol. 2013 Jan 1;7(1):1-3. doi: 10.1177/193229681300700101. No abstract available. PMID 23439154
- [Background] Kovatchev BP, Patek SD, Ortiz EA, Breton MD. Assessing sensor accuracy for non-adjunct use of continuous glucose monitoring. Diabetes Technol Ther. 2015 Mar;17(3):177-86. doi: 10.1089/dia.2014.0272. Epub 2014 Dec 1. PMID 25436913
- [Background] Bailey TS, Chang A, Christiansen M. Clinical accuracy of a continuous glucose monitoring system with an advanced algorithm. J Diabetes Sci Technol. 2015 Mar;9(2):209-14. doi: 10.1177/1932296814559746. Epub 2014 Nov 3. PMID 25370149
- [Background] Allen NA, Jacelon CS, Chipkin SR. Feasibility and acceptability of continuous glucose monitoring and accelerometer technology in exercising individuals with type 2 diabetes. J Clin Nurs. 2009 Feb;18(3):373-83. doi: 10.1111/j.1365-2702.2008.02533.x. PMID 19191984
- [Background] Allen NA, Fain JA, Braun B, Chipkin SR. Continuous glucose monitoring counseling improves physical activity behaviors of individuals with type 2 diabetes: A randomized clinical trial. Diabetes Res Clin Pract. 2008 Jun;80(3):371-9. doi: 10.1016/j.diabres.2008.01.006. Epub 2008 Mar 4. PMID 18304674
- [Background] Vigersky RA, Fonda SJ, Chellappa M, Walker MS, Ehrhardt NM. Short- and long-term effects of real-time continuous glucose monitoring in patients with type 2 diabetes. Diabetes Care. 2012 Jan;35(1):32-8. doi: 10.2337/dc11-1438. Epub 2011 Nov 18. PMID 22100963
- [Background] Fonda SJ, Salkind SJ, Walker MS, Chellappa M, Ehrhardt N, Vigersky RA. Heterogeneity of responses to real-time continuous glucose monitoring (RT-CGM) in patients with type 2 diabetes and its implications for application. Diabetes Care. 2013 Apr;36(4):786-92. doi: 10.2337/dc12-1225. Epub 2012 Nov 19. PMID 23172975
- [Background] Cox DJ, Tisdelle DA, Culbert JP. Increasing adherence to behavioral homework assignments. J Behav Med. 1988 Oct;11(5):519-22. doi: 10.1007/BF00844844. PMID 3236383
- [Background] Cox DJ, Taylor AG, Nowacek G, Holley-Wilcox P, Pohl SL, Guthrow E. The relationship between psychological stress and insulin-dependent diabetic blood glucose control: preliminary investigations. Health Psychol. 1984;3(1):63-75. doi: 10.1037//0278-6133.3.1.63. PMID 6536483
- [Background] Cox D, Gonder-Frederick L, McCall A, Kovatchev B, Clarke W. The effects of glucose fluctuation on cognitive function and QOL: the functional costs of hypoglycaemia and hyperglycaemia among adults with type 1 or type 2 diabetes. Int J Clin Pract Suppl. 2002 Jul;(129):20-6. PMID 12166601
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr; American Diabetes Association. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2013 Nov;36(11):3821-42. doi: 10.2337/dc13-2042. Epub 2013 Oct 9. PMID 24107659
- [Background] Anderson RM, Funnell MM, Fitzgerald JT, Marrero DG. The Diabetes Empowerment Scale: a measure of psychosocial self-efficacy. Diabetes Care. 2000 Jun;23(6):739-43. doi: 10.2337/diacare.23.6.739. PMID 10840988
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] McGuire BE, Morrison TG, Hermanns N, Skovlund S, Eldrup E, Gagliardino J, Kokoszka A, Matthews D, Pibernik-Okanovic M, Rodriguez-Saldana J, de Wit M, Snoek FJ. Short-form measures of diabetes-related emotional distress: the Problem Areas in Diabetes Scale (PAID)-5 and PAID-1. Diabetologia. 2010 Jan;53(1):66-9. doi: 10.1007/s00125-009-1559-5. Epub 2009 Oct 20. PMID 19841892
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Camarri B, Eastwood PR, Cecins NM, Thompson PJ, Jenkins S. Six minute walk distance in healthy subjects aged 55-75 years. Respir Med. 2006 Apr;100(4):658-65. doi: 10.1016/j.rmed.2005.08.003. Epub 2005 Oct 17. PMID 16229997
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Goff DC Jr, Lloyd-Jones DM, Smith SC Jr, Blum C, Schwartz JS; 2013 ACC/AHA Cholesterol Guideline Panel. Treatment of blood cholesterol to reduce atherosclerotic cardiovascular disease risk in adults: synopsis of the 2013 American College of Cardiology/American Heart Association cholesterol guideline. Ann Intern Med. 2014 Mar 4;160(5):339-43. doi: 10.7326/M14-0126. PMID 24474185
- [Background] Mayer SB, Jeffreys AS, Olsen MK, McDuffie JR, Feinglos MN, Yancy WS Jr. Two diets with different haemoglobin A1c and antiglycaemic medication effects despite similar weight loss in type 2 diabetes. Diabetes Obes Metab. 2014 Jan;16(1):90-3. doi: 10.1111/dom.12191. Epub 2013 Aug 29. PMID 23911112
- [Background] Oldroyd J, Banerjee M, Heald A, Cruickshank K. Diabetes and ethnic minorities. Postgrad Med J. 2005 Aug;81(958):486-90. doi: 10.1136/pgmj.2004.029124. PMID 16085737
- [Background] Cox DJ, Taylor AG, Singh H, Moncrief M, Diamond A, Yancy WS Jr, Hegde S, McCall AL. Glycemic load, exercise, and monitoring blood glucose (GEM): A paradigm shift in the treatment of type 2 diabetes mellitus. Diabetes Res Clin Pract. 2016 Jan;111:28-35. doi: 10.1016/j.diabres.2015.10.021. Epub 2015 Oct 21. PMID 26556234
- [Background] Cox DJ, Taylor AG, Moncrief M, Diamond A, Yancy WS Jr, Hegde S, McCall AL. Continuous Glucose Monitoring in the Self-management of Type 2 Diabetes: A Paradigm Shift. Diabetes Care. 2016 May;39(5):e71-3. doi: 10.2337/dc15-2836. Epub 2016 Mar 17. No abstract available. PMID 26989181
- [Background] Brunk DR, Taylor AG, Clark ML, Williams IC, Cox DJ. A Culturally Appropriate Self-Management Program for Hispanic Adults With Type 2 Diabetes and Low Health Literacy Skills. J Transcult Nurs. 2017 Mar;28(2):187-194. doi: 10.1177/1043659615613418. Epub 2016 Jul 9. PMID 26525585
- [Background] Farmer AJ, Perera R, Ward A, Heneghan C, Oke J, Barnett AH, Davidson MB, Guerci B, Coates V, Schwedes U, O'Malley S. Meta-analysis of individual patient data in randomised trials of self monitoring of blood glucose in people with non-insulin treated type 2 diabetes. BMJ. 2012 Feb 27;344:e486. doi: 10.1136/bmj.e486. PMID 22371867
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Hinderliter AL, Sherwood A, Craighead LW, Lin PH, Watkins L, Babyak MA, Blumenthal JA. The long-term effects of lifestyle change on blood pressure: One-year follow-up of the ENCORE study. Am J Hypertens. 2014 May;27(5):734-41. doi: 10.1093/ajh/hpt183. Epub 2013 Oct 1. PMID 24084586
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Miller CK, Kristeller JL, Headings A, Nagaraja H. Comparison of a mindful eating intervention to a diabetes self-management intervention among adults with type 2 diabetes: a randomized controlled trial. Health Educ Behav. 2014 Apr;41(2):145-54. doi: 10.1177/1090198113493092. Epub 2013 Jul 12. PMID 23855018
- [Background] Ekong G, Kavookjian J. Motivational interviewing and outcomes in adults with type 2 diabetes: A systematic review. Patient Educ Couns. 2016 Jun;99(6):944-52. doi: 10.1016/j.pec.2015.11.022. Epub 2015 Dec 4. PMID 26699083
- [Background] Foster-Powell K, Holt SH, Brand-Miller JC. International table of glycemic index and glycemic load values: 2002. Am J Clin Nutr. 2002 Jul;76(1):5-56. doi: 10.1093/ajcn/76.1.5. PMID 12081815
- [Background] Parkin CG, Buskirk A, Hinnen DA, Axel-Schweitzer M. Results that matter: structured vs. unstructured self-monitoring of blood glucose in type 2 diabetes. Diabetes Res Clin Pract. 2012 Jul;97(1):6-15. doi: 10.1016/j.diabres.2012.03.002. Epub 2012 Mar 30. PMID 22464874
- [Background] Polonsky WH, Fisher L. Self-monitoring of blood glucose in noninsulin-using type 2 diabetic patients: right answer, but wrong question: self-monitoring of blood glucose can be clinically valuable for noninsulin users. Diabetes Care. 2013 Jan;36(1):179-82. doi: 10.2337/dc12-0731. PMID 23264290
- [Background] Tsalatsanis A, Gil-Herrera E, Yalcin A, Djulbegovic B, Barnes L. Designing patient-centric applications for chronic disease management. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:3146-9. doi: 10.1109/IEMBS.2011.6090858. PMID 22255007
- [Background] Cox DJ, Gonder-Frederick L, Polonsky W, Schlundt D, Kovatchev B, Clarke W. Blood glucose awareness training (BGAT-2): long-term benefits. Diabetes Care. 2001 Apr;24(4):637-42. doi: 10.2337/diacare.24.4.637. PMID 11315822
- [Background] Cox D, Ritterband L, Magee J, Clarke W, Gonder-Frederick L. Blood glucose awareness training delivered over the internet. Diabetes Care. 2008 Aug;31(8):1527-8. doi: 10.2337/dc07-1956. Epub 2008 May 13. PMID 18477813
- [Background] Jilcott S, Ammerman A, Sommers J, Glasgow RE. Applying the RE-AIM framework to assess the public health impact of policy change. Ann Behav Med. 2007 Oct;34(2):105-14. doi: 10.1007/BF02872666. PMID 17927550
- [Background] Augustin LSA, Kendall CWC, Jenkins DJA, Willett WC, Astrup A, Barclay AW, Bjorck I, Brand-Miller JC, Brighenti F, Buyken AE, Ceriello A, La Vecchia C, Livesey G, Liu S, Riccardi G, Rizkalla SW, Sievenpiper JL, Trichopoulou A, Wolever TMS, Baer-Sinnott S, Poli A. Glycemic index, glycemic load and glycemic response: An International Scientific Consensus Summit from the International Carbohydrate Quality Consortium (ICQC). Nutr Metab Cardiovasc Dis. 2015 Sep;25(9):795-815. doi: 10.1016/j.numecd.2015.05.005. Epub 2015 May 16. PMID 26160327
- [Background] Greaves CJ, Sheppard KE, Abraham C, Hardeman W, Roden M, Evans PH, Schwarz P; IMAGE Study Group. Systematic review of reviews of intervention components associated with increased effectiveness in dietary and physical activity interventions. BMC Public Health. 2011 Feb 18;11:119. doi: 10.1186/1471-2458-11-119. PMID 21333011
- [Background] Runchey SS, Pollak MN, Valsta LM, Coronado GD, Schwarz Y, Breymeyer KL, Wang C, Wang CY, Lampe JW, Neuhouser ML. Glycemic load effect on fasting and post-prandial serum glucose, insulin, IGF-1 and IGFBP-3 in a randomized, controlled feeding study. Eur J Clin Nutr. 2012 Oct;66(10):1146-52. doi: 10.1038/ejcn.2012.107. Epub 2012 Aug 15. PMID 22892437
- [Background] Liu AG, Most MM, Brashear MM, Johnson WD, Cefalu WT, Greenway FL. Reducing the glycemic index or carbohydrate content of mixed meals reduces postprandial glycemia and insulinemia over the entire day but does not affect satiety. Diabetes Care. 2012 Aug;35(8):1633-7. doi: 10.2337/dc12-0329. Epub 2012 Jun 11. PMID 22688548
- [Background] Colberg SR, Grieco CR, Somma CT. Exercise effects on postprandial glycemia, mood, and sympathovagal balance in type 2 diabetes. J Am Med Dir Assoc. 2014 Apr;15(4):261-6. doi: 10.1016/j.jamda.2013.11.026. Epub 2014 Feb 6. PMID 24508328
- [Background] Turcotte LP, Fisher JS. Skeletal muscle insulin resistance: roles of fatty acid metabolism and exercise. Phys Ther. 2008 Nov;88(11):1279-96. doi: 10.2522/ptj.20080018. Epub 2008 Sep 18. PMID 18801860
- [Background] Rynders CA, Weltman JY, Jiang B, Breton M, Patrie J, Barrett EJ, Weltman A. Effects of exercise intensity on postprandial improvement in glucose disposal and insulin sensitivity in prediabetic adults. J Clin Endocrinol Metab. 2014 Jan;99(1):220-8. doi: 10.1210/jc.2013-2687. Epub 2013 Dec 20. PMID 24243632
- [Background] Bosi E, Scavini M, Ceriello A, Cucinotta D, Tiengo A, Marino R, Bonizzoni E, Giorgino F; PRISMA Study Group. Intensive structured self-monitoring of blood glucose and glycemic control in noninsulin-treated type 2 diabetes: the PRISMA randomized trial. Diabetes Care. 2013 Oct;36(10):2887-94. doi: 10.2337/dc13-0092. Epub 2013 Jun 4. PMID 23735724

DOCUMENTS (1):
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03207893/ICF_000.pdf